CLINICAL TRIAL: NCT07058207
Title: Weight Management in Obese Cancer Patients During Curative Active Treatment (CANOBESE Study): A Feasibility Study
Brief Title: Weight Management in Obese Cancer Patients During Curative Active Treatment
Acronym: CANOBESE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: World Cancer Research Fund International (Other); Institut Català d'Oncologia (Other)
Responsible Party: Principal Investigator, Lorena Arribas, Principal Investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR079/25
Record Dates: First submitted 2025-06-10; First posted 2025-07-10 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Solid Neoplasm; Stage II-IV; Curative Treatment
Keywords: Obesity; Neoplasms; Antineoplasic agents; Chemotherapy; Radiotherapy; Weight Loss; Physical Activity; Feasibility Studies; Patient Compliance; Patient Motivation; Patient Adherence; Patient Dropouts; Treatment-related adverse effects; Biomarkers; nutritional intervention; curative-intent treatment
MeSH Terms: conditions — Obesity; Neoplasms; Weight Loss; Motor Activity; Patient Compliance; Patient Dropouts

STUDY DESIGN:
Intervention Model Description: Single-arm intervention study designed to assess feasibility, accrual rate, retention, compliance and safety of a multimodal weight management program in obese cancer patients undergoing curative treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients with obesity with active curative treatment (Experimental): Fifty adult cancer patients with obesity (BMI ≥30 kg/m²) newly diagnosed with stage II-IV solid tumors undergoing curative-intent treatment. Participants will receive a multimodal weight management program combining dietary intervention, physicial activity and behavioral support.
  Interventions: Behavioral: Multimodal weight management program

INTERVENTIONS:
Behavioral: Multimodal weight management program — This intervention consists of three components:
  * Nutritional Counseling:
    * A personalized hypocaloric and high-protein diet is prescribed, based on individual energy requirements with a 20% caloric reduction.
    * The protein intake target is 1.5 g/kg/day to promote fat loss while maintaining muscle mass.
  * Exercise Program
    * Home-based, supervised aerobic and resistance training sessions conducted 3 times per week.
    * Each 60-minute session includes: 5 minutes flexibility, 25 minutes aerobic training, 25 minutes resistance training, and 5 minutes balance exercises.
  * Behavioral Support
    * Patients receive training in problem-solving strategies, motivation, and emotional self-regulation to improve adherence to both dietary and exercise goals.
    * Health professionals delivering the intervention are trained in behavior change techniques by a clinical psychologist.

SUMMARY:
This is a feasibility study intervention to fifty cancer patients with obesity and with newly diagnosed stage II-IV solid tumors undergoing curative treatment recruited at the Catalan Institute of Oncology (ICO) in L'Hospitalet, Spain.

The investigators hypothesize that weight management during cancer treatment could enhance health outcomes for this population. The feasibility of a multimodal weight loss management program will be assesses, including a personalized hypocaloric and high-protein diet combined with a supervised exercise home-program and behavioural support.

DETAILED DESCRIPTION:
The single-arm intervention will consist of a multimodal weight management program, including a personalized hypocaloric and high-protein diet combined with a supervised exercise home-program and behavioural support. Hypocaloric diet will be individualized according to their energy requirements estimated and then applying a 20% caloric restriction. In order to reduce body weight and maintain muscle mass, a high-protein diet will be provided consisting of 1.5 g of protein/kg/day.

Participants will be provided with a 3-day food record (3-DFR) chart prior to their baseline visit. After a full nutritional evaluation, the dietitian will create a diet plan unique to the participant. For those participants struggling to attain their recommended intake or anticipating protein intake to be challenging, an oral whey powder supplement will be provided for the duration of the study. Additional approaches to overcoming dietary challenges will include information/resources on nutritional symptom management that can impact dietary intake and/or high-protein recipes.

The exercise program will be based on supervised aerobic and resistance exercise home-based training sessions 3 times/week. The sessions will be 60 minutes long and will include 5 minutes of flexibility, followed by 25 minutes of aerobic exercises, 25 minutes of resistance exercises, and 5 minutes of balance exercises. The physiotherapist will supervise the sessions and will provide monthly individual face-to-face counselling to assure adherence to the protocol. The investigators have designed an individualized exercise program that fits the current patient's clinical situation. Each patient will receive a fitness tracker band to monitor his/her activity.

Behavioural support will include problem-solving strategies and practical tools to facilitate participants' self-control on emotional eating or stress-driven behaviours. Targeted behaviour goals will be set. A psychologist will provide technical support and training to the dietitian and the physiotherapist to improve their skills to provide behavioural changes and motivation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18+) with pathologically confirmed malignant solid tumors, stage II-IV, elected for oncological treatment (chemo, radio, or both) with curative intend.
* Expected oncological treatment time ≥ 3 months.
* BMI ≥ 30 kg/m²
* Resident in the Barcelona area up to the completion of cancer treatment.
* ECOG Perfomance Status (PS) 0-1
* Availability of internet access.

Exclusion Criteria:

* Patients with melanoma and brain tumours.
* Surgery as the only treatment.
* Tumour localizations with high risk of malnutrition (such as head and neck, upper gastrointestinal tract, or pancreatic cancer):
* Pregnancy or breastfeeding
* Another active malignancy
* Current health or medical condition that affects weight status, e.g., untreated hyper- or hypothyroidism,etc
* Pre-existing medical condition that precludes adherence to unsupervised exercise, e.g., severe orthopedic conditions, scheduled for a hip or knee replacement, bone metastases, paralysis, dementia, untreated stage 3 hypertension, or unstable angina, heart attack, congestive heart failure or conditions that dictated hospitalization or oxygen within 6-months.
* Unable to read or understand Spanish or Catalan
* Enrolled in a weight loss program
* Active suicidal ideation, anorexia, bulimia, binge eating disorder, current substance abuse or dependence (besides nicotine dependence)
* Use of pacemaker or another electrical implanted device
* History of bariatric (or LapBand) surgery, or considering or currently on a wait-list for bariatric or LapBand surgery
* Patients with any concurrent medical or psychological condition that, in the investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Accrual | From baseline to end of cancer treatment (3 to 9 months)
  Feasibility will be evaluated based on participant accrual, measured by the weekly enrollment rate and the total duration required to achieve the target sample size.
Retention | From baseline to end of cancer treatment (3 to 9 months)
  Feasibility will be assessed based on participant retention, monitored through attendance records signed at each visit. Investigators will calculate the retention rate, dropout rate, time to dropout, and reasons for discontinuation.
Fidelity of the programme delivery | From baseline to end of cancer treatment (3 to 9 months)
  Feasibility based on fidelity of the intervention will be assessed using a patient-completed checklist after each dietetic and physiotherapy session. Items will be scored as: +1: session content delivered as intended, 0: content omitted, -1: content delivered in a way that deviates from protocol.
  Fidelity scores will be aggregated, and if overall fidelity drops below 80%, retraining may be considered. Additionally, patients will complete a final evaluation form at the end of the program assessing intervention load, frequency, delivery format, behavioral support, and perceived value (e.g., effort, satisfaction, willingness to repeat).
Nutritional adherence | From baseline to end of cancer treatment (3 to 9 months)
  Feasibility based on adherence will be evaluated using a 24-hour dietary recall to assess energy and protein intake. At the end of the intervention period, dietary adherence will also be defined as a 10-20% reduction in baseline calorie intake, along with maintenance or an increase in protein intake.
Physical activity adherence | From baseline to end of cancer treatment (3 to 9 months)
  Feasibility based on physical activity adherence will be assessed through physiotherapist evaluations and wearable device tracking.
Ocurrance of any serious or life-threatening adverse events (Safety) | Throughout the study period (from baseline to end of intervention, 3 to 9 months)
  Safety will be evaluated by monitoring the occurrence of any serious or life-threatening adverse events that may be attributable to the intervention. Specifically, investigators will record physical or cardiac events resulting in overnight hospitalization. The clinical team will assess and document whether each event is related to the dietary, exercise, or behavioral components of the intervention.

SECONDARY OUTCOMES:
Change in Body Weight and Body Composition | Baseline to end of treatment (approx. 3 to 9 months)
  Assessed by bioelectrical impedance analysis (BIA, InBody S10) at each dietetic visit. Measures include total weight change (kg), fat mass (kg), and preservation of muscle mass. In patients with available imaging, body composition will be analyzed using CT scan at the L3 vertebral level.
Change in Eating Self-Efficacy | Baseline to the end of intervention (approx. 3 to 9 months)
  Eating self-efficacy will be assessed using the scenario-based Dieting Self-Efficacy Scale (DIET-SE), consisting of 11 items evaluating confidence in managing challenges to dietary self-control. Responses to each item are assessed on a Likert-type rating scale ranging from 0 (not at all confident) to 4 (very con-fident).
Change in physical activity self-efficacy | Baseline to the end of intervention (approx. 3 to 9 months)
  Exercise self-efficacy will be assessed using the modified Physical Activity Self-Efficacy Scale. A five-point Likert scale ranging from not at all confident (1) to very confident (5) will be used, higher scores indicating greater self-efficacy. Assessments will be conducted at baseline and at the end of the intervention.
Change in Autonomous Motivation | Baseline to the end of intervention (approx. 3 to 9 months)
  Autonomous motivation will be assessed using an adapted and abbreviated version of the Treatment Self-Regulation Questionnaire (TSRQ). This scale includes four items rated on a 5-point Likert scale ranging from 1 ("not at all true") to 5 ("very true"). Higher scores indicate greater autonomous motivation toward behavior change. One-to-one psychological support may be offered to participants with low scores to enhance engagement.
Modified Glasgow Prognostic Score | Baseline and end of treatment (3 to 9 months)
  Serum albumin and C-reactive protein levels will be used to calculate the Modified Glasgow Prognostic Score (mGPS) as a measure of systemic inflammation. Blood samples will be collected at baseline and at the end of the intervention, coinciding with routine clinical assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Arribas, PhD, MsC, RD, Principal Investigator — Catalan Institute of Oncology (ICO-Hospitalet). Bellvitge Biomedical Research Institute (IDIBELL)
Locations (1):
- Institut Català d'Oncologia. Catalan Institute of Oncology, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No